CLINICAL TRIAL: NCT04709224
Title: An Open-label Study to Determine the Pharmacokinetics, Safety and Tolerability of Single Ascending Doses of a Subcutaneous Injection of Lumateperone Long-Acting Injectable (LAI) Formulation in Patients With Schizophrenia
Brief Title: Pharmacokinetics, Safety, and Tolerability of Lumateperone Long-Acting Injectable in Patients With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Intra-Cellular Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ITI-007-025
Record Dates: First submitted 2020-12-29; First posted 2021-01-14 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: LAI Lumateperone 50 mg SC in the abdomen (Experimental)
  Interventions: Drug: Lumateperone Long-Acting Injectable
- Cohort 2: LAI Lumateperone 100 mg SC in the abdomen (Experimental)
  Interventions: Drug: Lumateperone Long-Acting Injectable
- Cohort 3: LAI Lumateperone 200 mg SC in the abdomen (Experimental)
  Interventions: Drug: Lumateperone Long-Acting Injectable
- Cohort 4: LAI Lumateperone 100 or 200 mg SC in the outer area of the upper arm (Experimental)
  Interventions: Drug: Lumateperone Long-Acting Injectable

INTERVENTIONS:
Drug: Lumateperone Long-Acting Injectable — Lumateperone Long-Acting Injectable

SUMMARY:
This is an open-label study to determine the pharmacokinetics, safety and tolerability of single ascending doses of lumateperone long-acting injectable formulation in patients with schizophrenia. Patients will be enrolled in one of up to four cohorts. All patients will receive oral lumateperone for 5 days, followed by a 5-day washout of oral lumateperone, then followed by a single dose of lumateperone LAI.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female patients aged 18 to 50 years, inclusive
* Clinical diagnosis of schizophrenia according to Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)
* Clinically stable and free from acute exacerbation of psychosis for at least 3 months prior to Screening per Investigator assessment
* On a stable dose of antipsychotic medication, including lumateperone, for at least 3 months prior to the Screening Visit
* Clinical Global Impression - Severity (CGI-S) score ≤ 3

Key Exclusion Criteria:

* Clinically significant abnormality within 2 years of Screening that, in the Investigator's opinion, may place the patient at risk or interfere with study outcome variables
* History of psychiatric condition other than schizophrenia that, in the Investigator's opinion, may be detrimental to participation in the study
* Any suicidal ideation within the 6 months prior to Screening, any suicidal behavior within 2 years prior to Screening based on the Columbia-Suicide Severity Rating Scale (C-SSRS) (excluding self-injurious, non-suicidal behavior), and/or Investigator assessment that the patient is a safety risk to him/herself or others
* Surgical or medical condition (active or chronic) that in the Investigator's opinion may interfere with drug absorption, distribution, metabolism, or excretion of the study drug or any other condition that may place the patient at risk; history of gastric bypass or sleeve gastrectomy; history of severe dystonic reaction on antipsychotics such as laryngeal spasm

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-05-23 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: Maximum observed plasma concentration (Cmax) of lumateperone and metabolites | predose and at multiple timepoints up to 7 weeks postdose
Pharmacokinetics: Time of maximum observed plasma concentration (Tmax) of lumateperone and metabolites | predose and at multiple timepoints up to 7 weeks postdose
Pharmacokinetics: Area under the plasma concentration-time curve from time zero to the last measurable concentration (AUC0-t) of lumateperone and metabolites | predose and at multiple timepoints up to 7 weeks postdose
Pharmacokinetics: Area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC0-inf) of lumateperone and metabolites | predose and at multiple timepoints up to 7 weeks postdose
Pharmacokinetics: Terminal elimination half-life (T1/2) of lumateperone and metabolites | predose and at multiple timepoints up to 7 weeks postdose
Pharmacokinetics: Maximum observed plasma concentration (Cmax,BR) of lumateperone and metabolites during burst-release phase | predose and at multiple timepoints up to 7 weeks postdose
Pharmacokinetics: Time of maximum observed plasma concentration (Tmax,BR) of lumateperone and metabolites during burst-release phase | predose and at multiple timepoints up to 7 weeks postdose
Pharmacokinetics: Area under the plasma concentration-time curve (AUC0-t,BR) of lumateperone and metabolites during burst-release phase | predose and at multiple timepoints up to 7 weeks postdose
Pharmacokinetics: Maximum observed plasma concentration (Cmax,SR) of lumateperone and metabolites during sustained-release phase | predose and at multiple timepoints up to 7 weeks postdose
Pharmacokinetics: Time of maximum observed plasma concentration (Tmax,SR) of lumateperone and metabolites during sustained-release phase | predose and at multiple timepoints up to 7 weeks postdose
Pharmacokinetics: Area under the plasma concentration-time curve (AUC0-t,SR) of lumateperone and metabolites during sustained-release phase | predose and at multiple timepoints up to 7 weeks postdose

SECONDARY OUTCOMES:
Percentage of participants with treatment-emergent AEs | up to 7 weeks postdose
Change from baseline in Systolic and Diastolic Blood Pressure | up to 7 weeks postdose
Change from baseline in hemoglobin | up to 7 weeks postdose
Change from baseline in platelet count | up to 7 weeks postdose
Change from baseline in white blood cell count | up to 7 weeks postdose
Change from baseline in aspartate aminotransferase | up to 7 weeks postdose
Change from baseline in alanine aminotransferase | up to 7 weeks postdose
Change from baseline in glucose | up to 7 weeks postdose
Change from baseline in creatine kinase | up to 7 weeks postdose
Change from baseline in ECG QT Interval | up to 7 weeks postdose
Change from baseline in Abnormal Involuntary Movement Scale | up to 7 weeks postdose
  AIMS is a measure of facial and oral movements, extremity movements and trunk movements. Items are rated on a scale from none (0) to severe (4).

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Clinical Site, Long Beach, California
  - Clinical Site, Marlton, New Jersey

IPD SHARING:
Plan to Share IPD: No